CLINICAL TRIAL: NCT02076932
Title: A Training Intervention Study in Late Pre- and Early Postmenopausal Women Investigating the Changes in Adipose Tissue Metabolism and Peripheral Insulin Sensitivity
Brief Title: Effects of Physical Training on Adipose Tissue Metabolism and Insulin Sensitivity in the Menopausal Transition Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other); Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Bente Merete Stallknecht, Professor, MD, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CWS menopause, adipose tissue
Record Dates: First submitted 2014-02-24; First posted 2014-03-04 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Menopause; Insulin Resistance; Body Composition, Beneficial
MeSH Terms: conditions — Insulin Resistance; Glucocorticoid Receptor Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Premenopausal women (Active Comparator): The premenopausal women will be attending Spinning classes.
  Interventions: Behavioral: Spinning
- Postmenopausal Women (Experimental): The postmenopausal women will be attending Spinning classes.
  Interventions: Behavioral: Spinning

INTERVENTIONS:
Behavioral: Spinning — After the baseline studies, the women will perform Spinning three times a week. Two of the sessions are performed on our location by trained instructors and the third training is self-training in a local fitness center where we provide free membership. All trainings are heart rate monitored.

SUMMARY:
The purpose of this study is to determine if physical exercise reduces the adverse changes in adipose tissue metabolism and insulin sensitivity that occurs in women during the menopausal transition.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal OR Postmenopausal (45-57 years)
* No chronical Diseases
* BMI > 18,5 and < 30
* Sedentary (no regular physical activity the last 2 years)
* Either regular bleeding (premenopausal) OR no menstruation for at least 2 years (postmenopausal)
* Plasma measurements:

Premenopausal: estradiol > 0.20nmol/l, Follicle Stimulating Hormone < 22 IU/l and progesterone > 2.5 nmol/l Postmenopausal: estradiol < 0.20nmol/l, Follicle Stimulating Hormone > 22 IU/l and progesterone from 0.3-2.5 nmol/l

Exclusion Criteria:

* Smoking
* Excessive alcohol intake
* Regular medication including hormone replacement treatment

Ages: 45 Years to 57 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Insulin stimulated uptake of glucose in adipose tissue | Baseline and 3 months
  Measured by Positron Emission Tomography-Computed tomography (PET/CT)
Hyperinsulinemic euglycemic clamp | Baseline and 3 months
  Glucose metabolized (mg/kg/min)
Adipose tissue distribution | Baseline and 3 months
  Accessed by Magnetic Resonance Imaging (MRI).

SECONDARY OUTCOMES:
Central insulin sensitivity | Baseline and 3 months
  Fasting plasma insulin, homeostasis model assessment insulin resistance and measures of central insulin sensitivity derived from an oral glucose tolerance test
Maximal oxygen uptake (ml/O2/kg/min) | Baseline and 3 months
  Measured using indirect calorimetry and an incremental bicycle protocol
Metabolic syndrome | Baseline and 3 months
  As measured by high density lipoprotein, triglycerides, waist circumference, blood pressure, mean arterial pressure, fasting glucose and composite metabolic syndrome scores
Health related quality of life | Baseline and 3 months
  Measured using questionaries, semi-structured interviews and observations
Anthropometry | Baseline and 3 months
  Measured using dual x-ray absorptiometry, height, weight, waist and hip circumference, sagittal abdominal height
Skeletal muscle biopsy | Baseline and 3 months
  Biochemical, proteomics, metabolomics, genomics and morphological analyses
Abdominal subcutaneous adipose tissue biopsy | Baseline and 3 months
  Biochemical, proteomics, metabolomics, genomics and morphological analyses
Resting metabolic rate | Baseline and 3 months
  Will be measured by indirect calorimetry
Physical activity level and duration of sleep | Baseline and 3 months
  Daily activity and duration of sleep will be recorded during one week using Actibelt® and self reporting
Microdialysis | Baseline and 3 months
  Adipose tissue microdialysis
Femoral subcutaneous adipose tissue biopsy | Baseline and 3 months
  Biochemical, proteomics, metabolomics, genomics and morphological analyses

OTHER OUTCOMES:
Dietary registration | Baseline and 3 months
  Daily food intake for three week days and one week-end day will be reported by the subjects

CONTACTS AND LOCATIONS:
Overall Officials: Ylva Hellsten, Proff., Principal Investigator — University of Copenhagen; Bente M Stallknecht, Proff. MD, Principal Investigator — University of Copenhagen
Locations (1):
- Department og Biomedical Sciences, Copenhagen N, Denmark